CLINICAL TRIAL: NCT05691816
Title: The Experience of the Child With Cancer When Port à Cath Needle : Child's Speech
Acronym: ELEAPort
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2022 USCLADE
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Pediatric Oncology
Keywords: Pediatrics; Cancer; Care; Experience; Port-a-cath
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This qualitative research refers to the descriptive phenomenological method of Hurssel which allows an analysis of the experience and an understanding of the phenomenon. Semi-structured interviews are carried out with 10 children followed for cancer in 3 pediatric hemato-oncology departments. The children interviewed are aged 6 to 12 and can be with their parents. A thematic analysis approach is used to analyze the data of this research.

ELIGIBILITY:
Inclusion Criteria:

* Child followed in pediatric oncology for cancer or hematological disease
* Child wearing a Port-a-cath needle placement and minimum use once a week

Exclusion Criteria:

* Child no speaking the French language

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6 to 12 with cancer and who have weekly care, requiring port-a-cath needle placement.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Experience of self management of port-a-cath needle placement | 60 minutes
  Evaluation from the patients' point of view on how they self-manage a port a cath needle placement, semi-structured qualitative interviews with patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Usclade, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France